CLINICAL TRIAL: NCT02104622
Title: Identify Training Strategies for Progressing Exoskeleton Users Towards Everyday Functional Ambulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, Arun Jayaraman, PT, PhD, Research Scientist, Shirley Ryan AbilityLab
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 89259
Record Dates: First submitted 2014-02-26; First posted 2014-04-04 (Estimated); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury; exoskeleton; ambulation; walking; robotics
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ReWalk training (Experimental)
  Interventions: Device: ReWalk Rehabilitation 2.0

INTERVENTIONS:
Device: ReWalk Rehabilitation 2.0

SUMMARY:
Many people with spinal cord injury are no longer able to walk and must use wheelchairs for mobility. These individuals experience greater rates of depression and lower quality of life. Many of these individuals express a strong desire to walk again, and report many psychosocial benefits to being eye to eye with peers in social interactions. Additionally, wheelchairs allow only limited community access, creating an additional obstacle to seeking out meaningful social roles in the community. Currently, there is new technology called robotic exoskeletons that would allow people with spinal cord injury to walk. These robotic exoskeletons also allow for curb, ramp, and stair negotiation, which are critical to community access. Current research has examined training with robotic exoskeletons indoors over level surfaces in clinical settings. This study will examine the potential for everyday use, including ramps, stairs, curbs and indoor and outdoor use.

ELIGIBILITY:
Inclusion Criteria:

* SCI level C6-8, T1-T12; L1-L5 incomplete or complete
* Be able to physically fit into the exoskeleton device;
* Be able to tolerate upright standing for a minimum of 30 minutes;
* Have sufficient upper body strength to use forearm crutches in standing and during ambulation (including full triceps strength and good hand function);
* Have hip, knee, and ankle range of motion within normal functional limits of walking;
* Have the ability to follow directions and demonstrate learning capacity;
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Cervical level SCI above C6
* History of severe osteoporosis;
* Weight above 220 pounds;
* Femur length above 47 cm or below 36 cm
* Joint contractures at the hip, knee, or ankle that limit normal range of motion (ROM) during ambulation;
* Cognitive and/or communication disability (e.g. due to brain injury);
* History of significant problems with skin break down or current skin break down;
* Any medical issue that precludes full weight bearing and ambulation (e.g. orthopedic injuries, pain, severe spasticity);
* Pregnancy;
* Cardiovascular conditions such as history of heart attack, high blood pressure, pacemaker, arrhythmia, heart failure, or stroke.

Ages: 12 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-02; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Change in 6 Minute Walk Test from baseline in distance, RPE and oxygen uptake | Session 1 (pre test, initial visit) and Session 20 (post test, between 6-8 weeks)
  The goal is to cover as much ground as possible over 6 minutes, the distance is measured with a measuring wheel. The instructions are "Walk continuously if possible, but do not be concerned if you need to slow down or stop to rest." At the end of 6 minutes the participant is asked to rate their exertion level on a Borg Scale of 6 - 20 points. The VO2 MAX data is collected during the test every 10 seconds
Change in 10 meter walk test from baseline in gait speed | Session 1 (pre test, initial visit) and Session 20 (post test, between 6-8 weeks)
  Measure the time in second for and individual to walk 10 meters. The test is Performed using a "flying start," patient walks 10 meters (33 ft) and the time is measured when the leading foot crosses the start line and the finish line. The instructions are: " Please walk this distance as fast as you safely can when I say go."
Time and assistive level to negotiate stairs, ramps, curbs, and turning. | Session 1 (pre test, initial visit) and Session 20 (post test, between 6-8 weeks)
Distance able to reach while standing and sitting | Session 1 (pre test, initial visit) and Session 20 (post test, between 6-8 weeks)

SECONDARY OUTCOMES:
Patient perception of Quality of Life | Session 1 (pre test, initial visit) and Session 20 (post test, between 6-8 weeks)
The Patient Health Questionnaire | Session 1 (pre test, initial visit) and Session 20 (post test, between 6-8 weeks)
  PHQ-9 is a 9-item self-report questionnaire designed to diagnose both the presence of depressive symptoms as well as to characterize the severity of depression. A single question rates how difficult problems have made it to do work, take care of things at home or get along with other people using a 4 level scale (not difficult at all to extremely difficult).
The Psychosocial Impact of Assistive Devices Scale | Session 1 (pre test, initial visit) and Session 20 (post test, between 6-8 weeks)
  The PIADS is a 26-item, self-report questionnaire designed to assess the effects of an assistive device on functional independence, well-being, and quality of life. The PIADS can be used to assess the impact of any assistive device (AD), prosthesis or medical procedure. It can be used to evaluate the impact of ADs over time and to match the devices with consumers. With its excellent psychometric properties, the PIADS fills a missing link in the assessment of ADs as well as in the examination of their acceptance and abandonment.
Activities-specific Balance Confidence Scale | Session 1 (pre test, initial visit) and Session 20 (post test, between 6-8 weeks)
Self reported Spinal Cord Independence Measure in activities of daily living | Session 1 (pre test, initial visit) and Session 20 (post test, between 6-8 weeks)
Pain measure by the Visual Analogue Scale | Session 1 (pre test, initial visit) and Session 20 (post test, between 6-8 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Arun Jayaraman, PT, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Rehabilitation Institute of Chicago, Chicago, Illinois, United States